CLINICAL TRIAL: NCT01292603
Title: An Adaptive, Comparative, Randomized, Parallel-group, Multi Center, Phase Ib Study of Subcutaneous (SC) Rituximab Versus Intravenous (IV) Rituximab Both in Combination With Chemotherapy (Fludarabine and Cyclophosphamide), in Patients With Previously Untreated CLL
Brief Title: A Study to Compare Subcutaneous Versus Intravenous MabThera (Rituximab) in Combination With Chemotherapy in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO25341; 2010-021380-32 (EudraCT Number)
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; Rituximab

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: rituximab [MabThera]
- 2 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: rituximab [MabThera]
- 3 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: rituximab [MabThera]

INTERVENTIONS:
Drug: Cyclophosphamide — Days 1-3 or Days 1-5 of cycles 1-6
Drug: Fludarabine — Days 1-3 or Days 1-5 of cycles 1-6
Drug: rituximab [MabThera] — One cycle of intravenous MabThera, followed by 5 cycles of subcutaneous MabThera
  Arms: 3
Drug: rituximab [MabThera] — After 4 cycles of intravenous MabThera without experiencing grade 3 or 4 infusion-related reactions. patients will receive 1 additional cycle of intravenous MabThera and 1 cycle of subcutaneous MabThera.
  Arms: 1
Drug: rituximab [MabThera] — 6 cycles of intravenous MabThera
  Arms: 2

SUMMARY:
This randomized, parallel-group, multi-center study will compare the pharmacokinetics and safety of subcutaneous administration of MabThera (rituximab) versus intravenous MabThera in combination with chemotherapy in previously untreated patients with chronic lymphocytic leukemia (CLL). The study consists of 2 parts. In part 1, patients who have previously received 4 cycles of intravenous MabThera will receive in Cycle 5 intravenous MabThera and in Cycle 6 subcutaneous MabThera. In part 2, patients will be randomized to receive either 6 cycles of intravenous MabThera, or 1 cycle of intravenous MabThera and 5 cycles of subcutaneous MabThera. Additionally, all patients will receive chemotherapy (fludarabine and cyclophosphamide) on Days 1-3 or Days 1-5 of every cycle. The anticipated time on study drug is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Patients with treatment-requiring chronic lymphocytic leukemia (CLL)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy >6 months

Exclusion Criteria:

* Transformation to aggressive B-cell malignancy
* History of other malignancy unless the patient was treated with curative intent and has been in remission for more than 5 years prior to enrolment
* HIV or Hepatitis B positive unless clearly due to vaccination
* Inadequate liver or renal function
* Any coexisting medical or psychological condition that would preclude participation in the required study procedures

Additional exclusion criterion for Part 1:

* Any previous treatment for CLL except for up to 4 cycles of rituximab IV in combination with FC chemotherapy as first-line treatment for CLL

Additional exclusion criterion for Part 2:

* Any previous treatment for CLL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-04-18 (Actual); Primary Completion 2014-05-07 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (84):
- Argentina (3):
  - Fundaleu; Haematology, Buenos Aires
  - Cemic; Haematology, Buenos Aires
  - HOSPITAL PRIVADO - CENTRO MEDICO DE CÓRDOBA; Dpto Oncología, Córdoba
- Australia (6):
  - St George Hospital; Department of Haematology, Kogarah, New South Wales
  - Royal Brisbane and Women'S Hospital; Haematology, Herston, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Queen Elizabeth Hospital; Haematology, Woodville South, South Australia
  - St Vincent'S Hospital; Haematology, Fitzroy, Victoria
  - Frankston Hospital; Oncology/Haematology, Frankston, Victoria
- Brazil (4):
  - Hospital da Cidade de Passo Fundo; Centro de Pesquisa em Oncologia, Passo Fundo, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Sirio Libanes; Centro de Oncologia, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Canada (4):
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - Centre de sante et de services sociaux Rimouski Neigette, Rimouski, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Chile (2):
  - Instituto Nacional del Cancer, Santiago
  - Centro Internacional de Estudios Clínicos (CIEC), Santiago
- Croatia (2):
  - Clinical Hospital Merkur; Dept of Haematology, Zagreb
  - University Hospital Center Zagreb; Haematology Department, Zagreb
- Czechia (3):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - University Hospital and Medical School; IV.Dept. of Internal Medicine and Hematology, Hradec Králové
  - Vseobecna Fakultni Nemocnice v Praze, I. Interni Klinika - Klinika Hematoonkologie VFN a 1. LF UK, Prague
- France (5):
  - Centre Francois Baclesse, Caen
  - Institut J Paolii Calmettes; Onco Hematologie 1, Marseille
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - Hopital Robert Debre; Hematologie Clinique, Reims
  - Hopitaux De Brabois; Hematologie Medecine Interne, Vandœuvre-lès-Nancy
- Germany (15):
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Onkologischer Schwerpunkt am Oskar-Helene-Heim; Dres. Herrenberger, Keitel-Wittig u. Kirsch, Berlin
  - Klinik der Uni zu Köln; Klinik für Innere Medizin, Cologne
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Klinikum Frankfurt; Medizinische Klinik I, Frankfurt (Oder)
  - Universitätsklinikum Greifswald Klinik für Innere Medizin C und Poliklinik, Greifswald
  - Onkologische Schwerpunktpraxis Dres. Bernd Gaede, Hans-Ulrich Ehlers, Ulrike Rodewig u.w., Hanover
  - Gemeinschaftspraxis Dr. Siehl & Dr. Soeling, Kassel
  - K&K Studien GbR, Landshut
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
  - Gemeinschaftspraxis Fr. Dr. med. Balser & Hr. Dr. med. Weidenbach, Marburg
  - Medizinisches Versorgungszentrum MOP, München
  - Klinikum Grosshadern der LMU, München
  - Gemeinschaftspraxis Dr. med. Holger Klaproth / Dr. med. Anca Astrid Cura, Neunkirchen/Saar
  - Prosper-Hospital, Medizinische Klinik I, Recklinghausen
- Greece (2):
  - Laiko General Hospital of Athens; A Propedeutical Clinic of Internal Medicine, Athens
  - Papageorgiou General Hospital of Thessaloniki; Hematology Clinic, Thessaloniki
- Italy (8):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Az. Osp. S. Maria Delle Croci; U.O. Di Ematologia, Ravenna, Emilia-Romagna
  - Ospedale Infermi Di Rimini; Unità Operativa di Oncologia e Oncoematologia, Rimini, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia; Clinica Ematologica, Udine, Friuli Venezia Giulia
  - Istituto S. Raffaele Monte Tabor; Divisione Ematologia E Utmo, Milan, Lombardy
  - ASST GRANDE OSPEDALE METROPOLITANO NIGUARDA; Struttura Complessa di Ematologia, Milan, Lombardy
  - Univ. Piemonte Est Amedeo Avogadro; Div.Ematologia- Dip.Clinica Med.Sperim.& Ircad, Novara, Piedmont
  - Policlinico G. B. Rossi; Divisione Di Ematologia, Verona, Veneto
- Mexico (3):
  - Centro Estatal De Cancerologia De Chihuahua; Servicio De Hematologia Banco De Sangre, Chihuahua City
  - Hospital General De Culiacan; Servicio De Hematologia, Culiacán
  - Hospital Universitario Dr. Jose E. Gonzalez; Haematology, Monterrey
- New Zealand (2):
  - Canterbury Health Laboratories; Haematology, Christchurch
  - Wellington Hospital; Wellington Blood and Cancer Centre, Newtown
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne; Klinika Hematologii i Transplantologii, Gdansk
  - Katedra i Klinika Hematoonkologii i Transplantacji Szpiku; Uniwersytetu Medycznego w Lublinie, Lublin
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie; Lymphoma Dept., Warsaw
  - Medical Uni of Wroclaw; Hematology, Wroclaw
- Portugal (2):
  - Hospital de Santa Maria; Servico de Hematologia e Transplantacao de Medula, Lisbon
  - IPO do Porto; Servico de Onco-Hematologia, Porto
- Russia (6):
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - City Clinical Hospital After Botkin; Hematology, Moscow
  - Haematology Research Center; Haematology, Moscow
  - Penza Regional Oncology Dispensary, Penza
  - Clinical MSCh No1, Perm
  - St. Petersburg State Medical University n.a. I.P. Pavlov; Hematology, transfusiology and transplanta, Saint Petersburg
- Slovakia (2):
  - National Oncology Inst. ; Dept. of Haematology, Bratislava
  - University Hospital; Clinic of Hematology & Transfusiology, Bratislava
- Spain (7):
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Universitario de la Princesa; Servicio de Hematologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Hematologia, Madrid
  - Hospital Clinico Universitario de Salamanca;Servicio de Hematologia, Salamanca
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Hematología, Toledo
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Turkey (Türkiye) (4):
  - Hacettepe Uni Medical Faculty; Hematology, Ankara
  - Istanbul University Cerrahpasa Medical Faculty; Hematology Department, Istanbul
  - Dokuz Eylul Uni ; Hematology, Izmir
  - Ege University ARGEFAR, Izmir

REFERENCES:
- [Derived] Assouline S, Buccheri V, Delmer A, Gaidano G, Trneny M, Berthillon N, Brewster M, Catalani O, Li S, McIntyre C, Sayyed P, Badoux X. Pharmacokinetics, safety, and efficacy of subcutaneous versus intravenous rituximab plus chemotherapy as treatment for chronic lymphocytic leukaemia (SAWYER): a phase 1b, open-label, randomised controlled non-inferiority trial. Lancet Haematol. 2016 Mar;3(3):e128-38. doi: 10.1016/S2352-3026(16)00004-1. PMID 26947201
- [Derived] Assouline S, Buccheri V, Delmer A, Gaidano G, McIntyre C, Brewster M, Catalani O, Hourcade-Potelleret F, Sayyed P, Badoux X. Pharmacokinetics and safety of subcutaneous rituximab plus fludarabine and cyclophosphamide for patients with chronic lymphocytic leukaemia. Br J Clin Pharmacol. 2015 Nov;80(5):1001-9. doi: 10.1111/bcp.12662. Epub 2015 Jul 29. PMID 25900065
- [Derived] Mao CP, Brovarney MR, Dabbagh K, Birnbock HF, Richter WF, Del Nagro CJ. Subcutaneous versus intravenous administration of rituximab: pharmacokinetics, CD20 target coverage and B-cell depletion in cynomolgus monkeys. PLoS One. 2013 Nov 12;8(11):e80533. doi: 10.1371/journal.pone.0080533. eCollection 2013. PMID 24265828
- [Derived] Shpilberg O, Jackisch C. Subcutaneous administration of rituximab (MabThera) and trastuzumab (Herceptin) using hyaluronidase. Br J Cancer. 2013 Sep 17;109(6):1556-61. doi: 10.1038/bjc.2013.371. Epub 2013 Sep 3. PMID 24002601

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part 1 a single dose of subcutaneous (SC) rituximab was administered at Cycle 6 to select a dose resulting in trough concentration (Ctrough) non-inferior to intravenous (IV) dose. In Part 2, participants were randomized to receive rituximab IV or SC, to demonstrate non-inferiority of rituximab Ctrough levels of SC dose compared with IV dose.
Groups:
- Part 1: Rituximab SC 1400 Milligrams (mg): Participant could have been enrolled any time during their treatment with rituximab IV in combination with fludarabine/cyclophosphamide (FC) prior to Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 milligrams per square meter (mg/m^2) on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 1: Rituximab SC 1600 mg: Participant could have been enrolled any time during their treatment with rituximab IV in combination with FC prior to Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1600 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 1: Rituximab SC 1870 mg: Participant could have been enrolled any time during their treatment with rituximab IV in combination with FC prior to Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1870 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 1: No SC Dose Received: These participants were withdrawn prior to SC treatment.
- Part 2 : Rituximab IV 500 mg/m^2: Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 0 Cycles 2-6: IV rituximab 500 mg/m^2 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 2: Rituximab SC 1600 mg: Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 0 Cycles 2-6: SC rituximab 1600 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Period: Part 1: Pilot Dose Selection Period
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: No SC Dose Received | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Started | 16 | 17 | 23 (1 participant received a dose of 1000mg of rituximab by oversight.) | 8 (These participants were withdrawn prior to SC treatment.) | 0 | 0
Completed | 16 | 17 | 23 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 8 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1: Regular Follow-Up Period
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: No SC Dose Received | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Started | 16 | 17 | 23 | 8 | 0 | 0
Completed | 10 (Participants withdrawn from regular follow-up who were still alive entered survival follow-up) | 10 (Participants withdrawn from regular follow-up who were still alive entered survival follow-up) | 17 (Participants withdrawn from regular follow-up who were still alive entered survival follow-up) | 7 | 0 | 0
Not Completed | 6 | 7 | 6 | 1 | 0 | 0
Not completed — Death | 3 | 1 | 3 | 1 | 0 | 0
Not completed — Disease Progression | 3 | 6 | 3 | 0 | 0 | 0
Period: Part 2: Dose Confirmation Period
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: No SC Dose Received | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Started | 0 | 0 | 0 | 0 | 88 | 88
Completed | 0 | 0 | 0 | 0 | 72 | 73
Not Completed | 0 | 0 | 0 | 0 | 16 | 15
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawn Prior to Treatment | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 7 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2
Period: Part 2: Regular Follow-Up
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: No SC Dose Received | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Started | 0 | 0 | 0 | 0 | 87 (Participants withdrawn from regular follow-up who were still alive entered survival follow-up) | 87 (Participants withdrawn from regular follow-up who were still alive entered survival follow-up)
Completed | 0 | 0 | 0 | 0 | 68 | 75
Not Completed | 0 | 0 | 0 | 0 | 19 | 12
Not completed — Death | 0 | 0 | 0 | 0 | 6 | 3
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 5 | 5
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 2
Period: Overall Survival Status
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: No SC Dose Received | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Started (Patients could enter survival follow-up directly after premature treatment withdrawal,) | 16 | 17 | 23 | 8 | 88 | 88
Completed (Overall survival.) | 13 | 16 | 20 | 7 | 72 | 78
Not Completed | 3 | 1 | 3 | 1 | 16 | 10
Not completed — Death | 3 | 1 | 3 | 1 | 16 | 10

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population (SAP): all participants who received at least one dose of study medication whether prematurely withdrawn or not. In Part 2 two participants randomized to the rituximab SC 1600 mg arm were included in Rituximab IV 500 mg/m^2 arm as they received only the first cycle of rituximab IV 375 mg/m^2.
Groups:
- Part 1: Rituximab SC 1400 Milligrams (mg): Participant could have been enrolled any time during their treatment with rituximab IV in combination with fludarabine/cyclophosphamide (FC) prior to Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Total: Total of all reporting groups
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg | Total
Number analyzed (Participants) | 16 | 17 | 22 | 89 | 85 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.13) | 60.4 (8.18) | 56.9 (6.79) | 58.7 (9.03) | 59.1 (8.87) | 58.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 7 | 36 | 25 | 76
  Male | 10 | 15 | 15 | 53 | 60 | 153

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Subcutaneous Rituximab Dose Resulting in Trough Concentration (Ctrough) Levels Non-Inferior to Intravenous Rituximab
Description: Ctrough is defined as the trough or minimum serum concentration. Pharmacokinetic parameters for rituximab were assessed during Cycles 5 (IV rituximab) and 6 (SC rituximab). Rituximab pharmacokinetic (PK) data from Part 1 were integrated into a population PK model using parametric, nonlinear, mixed-effects modelling. Rituximab IV 500 mg/m^2 administered once every 4 weeks was compared to fixed doses of rituximab SC between 1400 mg and 1870 mg. The dose selection was performed on Ctrough concentrations at Cycle 5 (pre-dose Cycle 6). A test of the probability of success was applied to each of the 100 replicates, and the percentage of replicates with a positive test corresponded to the probability of success of the trial.
Time Frame: Pre-dose and post-dose (15 minutes to end of infusion) on Day 1 and on Days 2, 5, 11 and 15 of Cycle 5 and Pre-dose, Post-dose on Days 2, 3, 5,11, 15 and 29 of Cycle 6; Pre-dose was taken 2 hours prior rituximab dose
Population: Enrolled (non-randomized) Pharmacokinetic Evaluable Population (Part 1) included all participants from Part 1 who did not significantly violate the inclusion or exclusion criteria, deviate significantly from the protocol or have unavailable or incomplete data which could influence the pharmacokinetic analysis.
Measure: Number; unit: mg
Groups:
- Part 1: Rituximab SC: Participant could have been enrolled any time during their treatment with rituximab IV in combination with FC prior to Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400, 1600 or 1870 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Arm/Group | Part 1: Rituximab SC
Number analyzed (Participants) | 56
mg | 1600

2. Primary Outcome: Part 2: Rituximab C Trough Levels at Cycle 5
Description: Ctrough is defined as the trough or minimum serum concentration in a given cycle of treatment. The objective of Part 2 was to demonstrate the comparability of the observed Ctrough of rituximab SC 1600 mg and rituximab IV 500 mg/m2 at Cycle 5, as assessed by a non-inferiority test with a lower boundary of at least 0.8 for the 90% CI.
Time Frame: +/- 25hours around the 28th day post the 5th Cycle of Rituximab administration
Population: Only participants who entered Part 2 of the study and had pharmacokinetic (PK) data available were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 69 | 65
μg/mL | 61.50 (89.54) | 97.53 (55.27)
Statistical Analysis 1: Comparison: Part 2 : Rituximab IV 500 mg/m^2 vs Part 2: Rituximab SC 1600 mg; Test type: Non-Inferiority or Equivalence — A standard non-inferiority margin of 0.8 for the ratio of Ctrough was used. The non-inferiority limit corresponds to a maximal 20 percent (%) loss in Ctrough which is considered acceptable given the high variability and range of Ctrough data, with an 80% power and a one-sided alpha of 0.05; Adjusted geometric mean ratio = 1.533, 90% CI 2-sided [1.269 to 1.852] — Ratio based on geometric scale and adjusted for the covariate tumor load at baseline

3. Secondary Outcome: Part 2: Observed Area Under the Serum Concentration-Curve (AUC) of Rituximab at Cycle 6
Description: AUC values were calculated by numerical integration using the linear trapezoidal rule. AUC levels were analyzed using the model below: Ln(AUC) = μ + τi + BlTLij + εij wherein, Ln is the natural log, μ denotes the overall mean effect, τi the effect in each treatment group, BlTLij the tumor load at baseline for each patient and εij a random error variable with normal distribution and mean 0. The treatment effect therein was based on a contrast statement in the model to calculate 90 % confidence intervals for ln(AUC SC)- ln(AUC IV).
Time Frame: Rituximab IV arm: pre-dose, post-dose and on Days 2, 3, 8 ,15, 29 of Cycle 6; Rituximab SC arm: pre-dose, and on Days 2, 3, 8 ,15, 29 of Cycle 6
Population: Only participants who entered Part 2 of the study and had PK data available were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 58 | 51
μg*day/mL | 3630.43 (38.61) | 4088.78 (37.52)
Statistical Analysis 1: Comparison: Part 2 : Rituximab IV 500 mg/m^2 vs Part 2: Rituximab SC 1600 mg; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.102, 90% CI 2-sided [0.979 to 1.242] — Ratio based on geometric scale and adjusted for the covariate tumor load at baseline

4. Secondary Outcome: Part 2: Maximum Observed Concentration (Cmax) of Rituximab at Cycle 6
Description: Cmax was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of time points of blood sampling and its measured concentration of rituximab in the blood samplings.
Time Frame: as for outcome 3
Population: Only participants who entered Part 2 of the study and had PK data available were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 58 | 51
μg/mL | 279.78 (23.96) | 202.16 (36.10)
Statistical Analysis 1: Comparison: Part 2 : Rituximab IV 500 mg/m^2 vs Part 2: Rituximab SC 1600 mg; Test type: Superiority or Other; Adjusted geometric mean ratio = 0.719, 90% CI 2-sided [0.653 to 0.792] — Ratio based on geometric scale and adjusted for the covariate tumor load at baseline

5. Secondary Outcome: Part 2: Time to Cmax (Tmax) of Rituximab at Cycle 6
Description: Multiple blood samples were obtained at pre-dose, post-dose and on Days 2, 3, 8 ,15, 29 of Cycle 6 in Rituximab IV arm, and at pre-dose, and on Days 2, 3, 8 ,15, 29 of Cycle 6 in Rituximab SC arm and time to peak plasma concentration of rituximab was determined.
Time Frame: as for outcome 3
Population: Only participants who entered Part 2 of the study and had PK data available were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 58 | 51
days | 0.22 (130.84) | 3.14 (87.62)
Statistical Analysis 1: Comparison: Part 2 : Rituximab IV 500 mg/m^2 vs Part 2: Rituximab SC 1600 mg; Test type: Superiority or Other; Adjusted geometric mean ratio = 14.884, 90% CI 2-sided [11.215 to 19.755] — Ratio based on geometric scale and adjusted for the covariate tumor load at baseline

6. Secondary Outcome: Part 2: Terminal Half-Life of Rituximab at Cycle 6
Description: The terminal half-life (t1/2) of rituximab is defined as the time required for the plasma concentration of rituximab to reach half of its original concentration.
Time Frame: as for outcome 3
Population: Only participants who entered Part 2 of the study and had PK data available were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 58 | 50
days | 30.09 (41.86) | 30.71 (33.19)
Statistical Analysis 1: Comparison: Part 2 : Rituximab IV 500 mg/m^2 vs Part 2: Rituximab SC 1600 mg; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.010, 90% CI 2-sided [0.895 to 1.139] — Ratio based on geometric scale and adjusted for the covariate tumor load at baseline

7. Secondary Outcome: Part 1: Percentage of Participants and Nurses Recording a Preference For Either SC or IV Administration
Description: In part 1 of the trial, upon completion of dosing in cycle 6, participants and their treating nurses were asked whether they have a preference of dosing route, IV vs SC
Time Frame: Days 4 to 5 in Cycle 6
Population: All participants in Part 1 were included in this analysis including 8 participants that did not receive SC rituximab.
Measure: Number; unit: percentage of participants or nurses
Groups:
- Part 1: Rituximab SC 1400 mg: Participant could have been enrolled any time during treatment with rituximab IV in combination with fludarabine/cyclophosphamide (FC) prior to Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 1: Rituximab SC 1600 mg: Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1600 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 1: Rituximab SC 1870 mg: Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1870 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Arm/Group | Part 1: Rituximab SC 1400 mg | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg
Number analyzed (Participants) | 16 | 17 | 23
percentage of participants or nurses
  Participants who preferred SC | 88.0 | 100.0 | 91.0
  Participants who preferred IV | 13.0 | 0.0 | 9.0
  Nurses who preferred SC | 88.0 | 100.0 | 91.0
  Nurses who preferred IV | 13.0 | 0.0 | 9.0

8. Secondary Outcome: Part 2: Physician/Nurse Opinion on Time Savings With Rituximab SC Compared With Rituximab IV
Description: Physicians and nurses who administered rituximab were asked to answer the following question: " If used in routine practice, on average, how much staff time could be saved with each administration of rituximab SC as compared to rituximab IV? (Please do not consider the time needed for the first IV administration, consider only the subsequent ones)". The number of nurses that responded for both the IV and SC arms was 70. The number of physicians that responded for the IV and SC arms were 78 and 81 respectively.
Time Frame: Days 4-5 in Cycle 6
Population: All the physicians and nurses who responded to the questionnaire were included in the analysis.
Measure: Number; unit: percentage of participants in the survey
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 78 | 81
percentage of participants in the survey
  Nurse: 4 or more hours | 21.0 | 21.0
  Nurse: At least 3 hours but less than 4 hours | 23.0 | 29.0
  Nurse: At least 2 hours but less than 3 hours | 26.0 | 23.0
  Nurse: At least 1 hour but less than 2 hours | 17.0 | 11.0
  Nurse: Less than 1 hour | 13.0 | 16.0
  Physician: 4 or more hours | 21.0 | 22.0
  Physician: At least 3 hours but less than 4 hours | 18.0 | 21.0
  Physician: At least 2 hours but less than 3 hours | 24.0 | 26.0
  Physician: At least 1 hour but less than 2 hours | 22.0 | 19.0
  Physician: Less than 1 hour | 10.0 | 7.0

9. Secondary Outcome: Part 2: Physician/Nurse Opinion on Convenience of Rituximab SC Compared With Rituximab IV
Description: Physicians and nurses who administered rituximab were asked to answer the following question: "Which formulation of rituximab (SC or IV) do you think is more convenient?" with pre-specified responses as below. Percentage of participants with specified answers were reported. The number of nurses that responded for both the IV and SC arms was 70. The number of physicians that responded for the IV and SC arms were 78 and 81 respectively.
Time Frame: Days 4-5 in Cycle 6
Population: All the physicians and nurses who responded to the questionnaire were included in the analysis.
Measure: Number; unit: percentage of participants in the survey
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 78 | 81
percentage of participants in the survey
  Nurse: Rituximab SC is much more convenient | 81.0 | 77.0
  Nurse: Rituximab SC is a little more convenient | 7.0 | 9.0
  Nurse: Both formulations are equally convenient | 9.0 | 4.0
  Nurse: Rituximab IV is a little more convenient | 3.0 | 10.0
  Nurse: Rituximab IV is much more convenient | 0.0 | 0.0
  Physician: Rituximab SC is much more convenient | 78.0 | 80.0
  Physician: Rituximab SC a little more convenient | 15.0 | 14.0
  Physician: Both formulations equally convenient | 6.0 | 6.0
  Physician: Rituximab IV a little more convenient | 0.0 | 0.0
  Physician: Rituximab IV is much more convenient | 0.0 | 0.0

10. Secondary Outcome: Part 1: Percentage of Participants With Anti-Rituximab Antibodies
Description: Blood samples for the assessment of antibodies against rituximab (HACAs) were drawn pre-dose at Cycle 5 and Cycle 6 in Part 1 and at each follow up visit until 24 months after the last dose.
Time Frame: Predose at Cycles 5 and 6 and at each follow up visit until 24 months after the last dose
Population: Safety Analysis Population (SAP): all participants who received at least one dose of study medication, whether prematurely withdrawn from the study or not. This included 8 participants that did not receive SC rituximab. n = number of participants analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Part 1: Rituximab SC: Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400, 1600 or 1870 mg on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Arm/Group | Part 1: Rituximab SC
Number analyzed (Participants) | 64
percentage of participants
  Pre-Dose Cycle 5: positive for HACAs (n=59) | 0.0
  Pre-Dose Cycle 5: negative for HACAs (n=59) | 100.0
  Post-Dose: positive for HACAs (n=61) | 5.0
  Post-Dose: negative for HACAs (n=61) | 95.1

11. Secondary Outcome: Part 2: Percentage of Participants With Anti-Rituximab Antibodies
Description: In Part 2, samples for the HACA assay were collected at each treatment cycle prior to the administration of rituximab and at each follow-up visit until 24 months after the last dose of rituximab.
Time Frame: Day 0 of Cycle 1 and Day 1 of Cycles 1, 2, 3, 4, 5, and 6 and at each follow-up visit until 24 months after the last dose of rituximab.
Population: SAP; n = number of participants analyzed for the specific parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 89 | 85
percentage of participants
  Baseline pre Cycle 1: positive for HACAs (n=87,85) | 0.0 | 2.4
  Baseline pre Cycle 1: negative for HACAs (n=87,85) | 100.0 | 97.6
  Post-Baseline: positive for HACAs (n=89,85) | 15.0 | 12.0
  Post-Baseline: negative for HACAs (n=89,85) | 85.0 | 88.0

12. Secondary Outcome: Part 1: Total Cluster Differentiation19 Positive (CD19+) B-Cell Counts by Visit
Description: CD 19 is a surface antigen (protein) present on B-lymphocytes.
Time Frame: Day 1 of Cycles 5 and 6 and Follow-up Days 28 and 56 and Follow-up Visits at Months 3, 6, 9, 12, 15,18, 21 and 24
Population: Part 1 SAP; n = number of participants analyzed at the specified visit.
Measure: Median (Full Range); unit: cells per microliter (cells/μL)
Groups:
- Part 1: Rituximab SC 1400 Milligrams (mg): Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Part 1: Rituximab SC 1000 mg: One participant enrolled in the rituximab SC 1870 mg subcohort received 1000 mg rituximab SC during Cycle 6 in error.
  Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1000 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Arm/Group | Part 1: Rituximab SC 1400 Milligrams (mg) | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: Rituximab SC 1000 mg | Part 1: No SC Dose Received
Number analyzed (Participants) | 16 | 17 | 22 | 1 | 8
cells per microliter (cells/μL)
  Cycle 5 Day 1 (n=15,13,19,1,2) | 2 [0 to 157] | 3 [0 to 419] | 0 [0 to 19] | 84 [NA to NA] — Only 1 participant was analyzed in this group. | 2 [1 to 2]
  Cycle 6 Day 1 (n=15,14,18,1,0) | 1 [0 to 90] | 2 [0 to 22] | 1 [0 to 5] | 27 [NA to NA] — Only 1 participant was analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 28 Day Visit (n=15,11,19,1,0) | 2 [0 to 113] | 2 [0 to 8] | 0 [0 to 7] | 7 [NA to NA] — Only 1 participant was analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 56 Day Visit (n=15,9,15,1,0) | 1 [0 to 215] | 3 [1 to 42] | 0 [0 to 2] | 14 [NA to NA] — Only 1 participant was analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 3 Month Visit (n=16,8,18,0,0) | 3 [0 to 469] | 1 [0 to 5] | 1 [0 to 6] | NA [NA to NA] — No participants were analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 6 Month Visit (n=15,13,17,1,0) | 2 [0 to 5929] | 1 [0 to 265] | 2 [0 to 96] | 51 [NA to NA] — Only 1 participant was analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 9 Month Visit (n=15,13,15,1,0) | 66 [0 to 15727] | 19 [1 to 728] | 29 [0 to 1153] | 74 [NA to NA] — Only 1 participant was analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 12 Month Visit (n=14,14,20,0,0) | 126 [4 to 1457] | 31 [0 to 2775] | 90 [2 to 1281] | NA [NA to NA] — No participants were analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 15 Month Visit (n=14,11,15,0,0) | 175 [14 to 2426] | 41 [3 to 6588] | 106 [29 to 500] | NA [NA to NA] — No participants were analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 18 Month Visit (n=13,14,15,0,0) | 175 [15 to 5871] | 82 [16 to 13749] | 189 [22 to 478] | NA [NA to NA] — No participants were analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 21 Month Visit (n=13,12,16,0,0) | 128 [27 to 10679] | 78 [9 to 314] | 149 [57 to 783] | NA [NA to NA] — No participants were analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.
  FU 24 Month Visit(n=12, 4,16,0,0) | 238 [29 to 11989] | 110 [25 to 2225] | 232 [69 to 1343] | NA [NA to NA] — No participants were analyzed in this group. | NA [NA to NA] — No participants were analyzed in this group.

13. Secondary Outcome: Part 1: Percentage of Participants With Total B-Cell Depletion by Visit
Description: Total B-cell depletion (normal B-cell plus Malignant B-cell depletion) was defined for each individual participant when the sum of CD5-/CD19+ (normal B-cells) and CD5+/CD19+ (malignant B-cells) cell counts decreased below 80 cells/μL.
Time Frame: Day 1 pre-dose of Cycles 5 and 6 and Follow-up Days 28 and 56 and Follow-up Visits at Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: Part 1 SAP; n = number of participants analyzed at the specified visit.
Measure: Number; unit: percentage of participants
Groups:
- Part 1: Rituximab SC 1400 mg: Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1400 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
- Rituximab SC 1000 mg: Participant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1000 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Arm/Group | Part 1: Rituximab SC 1400 mg | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Rituximab SC 1000 mg | Part 1: No SC Dose Received
Number analyzed (Participants) | 16 | 17 | 22 | 1 | 8
percentage of participants
  Cycle 5 Day 1 (n=15,1319,1,2) | 93.3 | 92.3 | 100.0 | 0.0 | 100.0
  Cycle 6 Day 1(n= 15,14,18,1,0) | 93.3 | 100.0 | 100.0 | 100.0 | NA — No participants were analyzed in this group.
  FU 28 Day Visit (n=15,11,19,1,0) | 93.3 | 100.0 | 100.0 | 100.0 | NA — No participants were analyzed in this group.
  FU 56 Day Visit (n=15,9,15,1,0) | 93.3 | 100.0 | 100.0 | 100.0 | NA — No participants were analyzed in this group.
  FU 3 Month Visit (n=16,8,18,0,0) | 93.8 | 100.0 | 100.0 | NA — No participants were analyzed in this group. | NA — No participants were analyzed in this group.
  FU 6 Month Visit (n=15,13,17,1,0) | 86.7 | 92.3 | 94.1 | 100.0 | NA — No participants were analyzed in this group.
  FU 9 Month Visit (n=15,13,15,1,0) | 53.3 | 84.6 | 60.0 | 100.0 | NA — No participants were analyzed in this group.
  FU 12 Month Visit (n=14,14,20,0,0) | 28.6 | 85.7 | 45.0 | NA — No participants were analyzed in this group. | NA — No participants were analyzed in this group.
  FU 15 Month Visit (n=14,11,15,0,0) | 35.7 | 54.5 | 40.0 | NA — No participants were analyzed in this group. | NA — No participants were analyzed in this group.
  FU 18 Month Visit (n=13,14,15,0,0) | 30.8 | 50.0 | 26.7 | NA — No participants were analyzed in this group. | NA — No participants were analyzed in this group.
  FU 21 Month Visit (n=13,12,16,0,0) | 30.8 | 50.0 | 18.8 | NA — No participants were analyzed in this group. | NA — No participants were analyzed in this group.
  FU 24 Month Visit (n=12,14,16,0,0) | 25.0 | 21.4 | 18.8 | NA — No participants were analyzed in this group. | NA — No participants were analyzed in this group.

14. Secondary Outcome: Part 2: Total CD19+ B-Cell Counts by Visit
Description: CD 19 is a surface antigen (protein) present on B-lymphocytes.
Time Frame: Cycle 1 pre-dose, 60 minutes post-dose, Days 2 and 3 in Cycle 2, day 1 pre-dose in Cycles 3, 4, 5 and 6, Follow-up Days 28 and 56, and Follow-up Visits at Months 3, 6, 9, 12, 15, and 18 and Withdrawal Visit
Population: Part 2 SAP; n = number of participants analyzed at the specified visit.
Measure: Median (Full Range); unit: cells/μL
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 89 | 85
cells/μL
  Cycle 1 - Baseline (n=80,80) | 68905 [3996 to 277645] | 50565 [640 to 453292]
  Cycle 2 - Pre-dose (n=71,74) | 338 [2 to 38252] | 253 [1 to 92469]
  Cycle 2 - Post-dose (n=65, 66) | 163 [3 to 13026] | 168 [1 to 32615]
  Cycle 2 Day 2 (n=54, 59) | 154 [6 to 10416] | 266 [0 to 40815]
  Cycle 2 Day 3 (n=48, 54) | 87 [0 to 14769] | 125 [0 to 13229]
  Cycle 3 Day 1 (n=67,68) | 12 [0 to 13118] | 8 [1 to 22392]
  Cycle 4 Day 1 (n=71,69) | 4 [0 to 17827] | 4 [0 to 18672]
  Cycle 5 Day 1 (n=68,67) | 2 [0 to 7146] | 2 [0 to 8542]
  Cycle 6 Day 1 (n=71,64) | 3 [0 to 3612] | 3 [0 to 4234]
  FU 28 Day Visit (n=66,64) | 2 [0 to 1299] | 2 [0 to 2749]
  FU 56 Day Visit (n=63,67) | 2 [0 to 14331] | 2 [0 to 3539]
  FU 3 Month Visit (n=67,67) | 2 [0 to 39037] | 2 [0 to 16413]
  FU 6 Month Visit (n=60,69) | 3 [0 to 1356] | 3 [0 to 22630]
  FU 9 Month Visit (n=65,64) | 35 [1 to 3776] | 30 [0 to 890]
  FU 12 Month Visit (n=60,61) | 91 [4 to 9372] | 104 [1 to 1770]
  FU 15 Month Visit (n=59,60) | 135 [6 to 16328] | 171 [5 to 9431]
  FU 18 Month Visit (n=57,58) | 134 [5 to 15404] | 223 [3 to 22363]
  FU 21 Month Visit (n=55,52) | 171 [5 to 7901] | 277 [5 to 39435]
  FU 24 Month Visit (n=56,51) | 214 [0 to 78010] | 256 [6 to 10482]
  Withdrawn/Termination (n=17,15) | 150 [2 to 90310] | 6 [0 to 35325]

15. Secondary Outcome: Part 2: Percentage of Participants With Total B-Cell Depletion by Visit
Description: as for outcome 13
Time Frame: Cycle 1 Pre-dose, 60 minutes post-dose, Days 2 and 3 in Cycle 2, day 1 in Cycles 3, 4, 5 and 6, Follow-up Days 28 and 56, and Follow-up Visits at Months 3, 6, 9, 12, 15, and 18 and Withdrawal Visit
Population: Part 2 SAP; n= number of participants analyzed at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Number analyzed (Participants) | 89 | 85
percentage of participants
  Cycle 1 - Baseline (n=80,80)) | 0.0 | 0.0
  Cycle 2 - Pre-dose (n=71, 74) | 23.9 | 31.1
  Cycle 2 - Post-dose (n=65, 66) | 32.3 | 37.9
  Cycle 2 Day 2 (n=54, 59) | 35.2 | 30.5
  Cycle 2 Day 3 (n=48, 54) | 50.0 | 37.0
  Cycle 3 Day 1 (n=67,68) | 73.1 | 76.5
  Cycle 4 Day 1 (n=71,69) | 83.1 | 84.1
  Cycle 5 Day 1 (n=68,67) | 88.2 | 89.6
  Cycle 6 Day 1 (n=71,64) | 95.8 | 95.3
  FU 28 Day Visit (n=66,64) | 95.5 | 96.9
  FU 56 Day Visit (n=63,67) | 92.1 | 97.0
  FU 3 Month Visit (n=67,67) | 95.5 | 92.5
  FU 6 Month Visit (n=60,69) | 88.3 | 91.3
  FU 9 Month Visit (n=65,64) | 66.2 | 70.3
  FU 12 Month Visit (n=60,61) | 43.3 | 42.6
  FU 15 Month Visit (n=59,60) | 33.9 | 30.0
  FU 18 Month Visit (n=57,58) | 24.6 | 25.9
  FU 21 Month Visit (n=55,52) | 14.5 | 19.2
  FU 24 Month Visit (n=56,51) | 10.7 | 15.7
  Withdrawn/Termination (n=17,15) | 41.2 | 73.3

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the time of initiation of treatment until 28 days after completion of study treatment in Cycle 6.
Description: New infections and all unrelated SAEs were reported until 9 months after the last dose of study treatment. All related SAEs were reported indefinitely. Secondary malignancies were reported until the end of the study or initiation of a new anti-leukemia treatment, whichever was earlier.
Groups:
- Part 1: Rituximab SC 1870 mg: PParticipant could have been enrolled any time during treatment with rituximab IV in combination with FC before Cycle 5. Participants received the following in 28-day cycles. Cycle 1: IV rituximab 375 mg/m^2 on Day 1 or Day 0 (according to local practice) Cycles 2-5: IV rituximab 500 mg/m^2 on Day 1 Cycle 6: SC rituximab 1870 on Day 1 Cycles 1-6: IV fludarabine 25 mg/m^2 on Days 1-3 (or as an oral dose of 24 mg/m^2 on Days 1-5 or 30-40 mg/m^2 on Days 1-3), and IV cyclophosphamide 250 mg/m^2 on Days 1-3 (or as an oral dose of 150 mg/m^2 on Days 1-5 or 200-250 mg/m^2 on Days 1-3).
Arm/Group | Part 1: Rituximab SC 1400 mg | Part 1: Rituximab SC 1600 mg | Part 1: Rituximab SC 1870 mg | Part 1: Rituximab SC 1000 mg | Part 1: No SC Dose Received | Part 2 : Rituximab IV 500 mg/m^2 | Part 2: Rituximab SC 1600 mg
Serious Adverse Events (participants affected / at risk) | 5/16 | 8/17 | 4/22 | 1/1 | 3/8 | 35/89 | 32/85
Other Adverse Events (participants affected / at risk) | 13/16 | 16/17 | 21/22 | 1/1 | 7/8 | 80/89 | 81/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Rituximab SC 1400 mg (N=16) | Part 1: Rituximab SC 1600 mg (N=17) | Part 1: Rituximab SC 1870 mg (N=22) | Part 1: Rituximab SC 1000 mg (N=1) | Part 1: No SC Dose Received (N=8) | Part 2 : Rituximab IV 500 mg/m^2 (N=89) | Part 2: Rituximab SC 1600 mg (N=85)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1 | 1 | 4 | 9
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic Retinal Oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound Dehiscene (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Guillain- Barre Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis Cryptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulpitis Dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meralgia Paraesthetica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash Maculo- Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
BARTHOLINITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3 | 1
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
REFRACTORY ANAEMIA WITH AN EXCESS OF BLASTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ENCEPHALITIS AUTOIMMUNE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Rituximab SC 1400 mg (N=16) | Part 1: Rituximab SC 1600 mg (N=17) | Part 1: Rituximab SC 1870 mg (N=22) | Part 1: Rituximab SC 1000 mg (N=1) | Part 1: No SC Dose Received (N=8) | Part 2 : Rituximab IV 500 mg/m^2 (N=89) | Part 2: Rituximab SC 1600 mg (N=85)
Neutropenia (Blood and lymphatic system disorders) | 7 | 8 | 9 | 1 | 3 | 51 | 54
Leukopenia (Blood and lymphatic system disorders) | 3 | 6 | 0 | 0 | 1 | 15 | 16
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 1 | 2 | 21 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 1 | 1 | 25 | 20
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 4 | 0 | 2 | 31 | 32
Vomiting (Gastrointestinal disorders) | 2 | 2 | 7 | 0 | 2 | 20 | 18
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 3 | 0 | 1 | 9 | 10
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 7 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 5 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 5 | 1 | 0 | 1 | 23 | 26
Chills (General disorders) | 1 | 3 | 1 | 0 | 1 | 9 | 12
Injection site pain (General disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 14
Injection site erythema (General disorders) | 0 | 2 | 4 | 0 | 0 | 0 | 22
Asthenia (General disorders) | 1 | 2 | 1 | 0 | 0 | 16 | 8
Fatigue (General disorders) | 0 | 3 | 0 | 0 | 1 | 9 | 9
Chest discomfort (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 4 | 0 | 0 | 5 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 13 | 10
Herpes zoster (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 5 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 7 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 8 | 7
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3 | 7
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 0 | 9 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 6 | 14
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 4 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 10 | 10
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 3 | 0 | 0 | 10 | 7
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 6 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 5
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 6 | 1
DYSCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Venous Disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.